CLINICAL TRIAL: NCT07309991
Title: Impact of Arterial Partial Pressure of Oxygen on Anastomotic Leakage After Esophagectomy
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yang Hong, Professor, Sun Yat-sen University
Other Study IDs: B2025-825-01
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Carcinoma; Esophageal Adenocarcinoma; Esophagectomy; PaO2; Esophageal Anastomotic Leakeage
Keywords: Effect of Postoperative PaO₂ on Anastomotic Leakage Following Esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Pa02 Group: Patients were defined as belonging to the Low PaO₂ group if they exhibited at least one recorded instance of PaO₂ <80 mmHg within the first postoperative week.
- Normal PaO2 Group: Patients maintained a PaO₂ ≥80 mmHg throughout the first postoperative week.

SUMMARY:
This study aims to determine whether postoperative hypoxia (arterial partial pressure of oxygen (PaO₂)<80 mmHg) is an independent risk factor for anastomotic leakage after esophagectomy. We conducted a retrospective analysis of cases from our center over the past five years, stratifying patients into Low Pa0₂ Group and Normal Pa0₂ Group based on postoperative oxygen levels and comparing the incidence of anastomotic leakage between the groups. The goal is to establish whether hypoxia is a causative risk factor and whether correcting it can reduce the risk of anastomotic leakage.

DETAILED DESCRIPTION:
This retrospective study included all patients who underwent radical esophagectomy at our center over the past five years. After screening based on inclusion and exclusion criteria, PaO₂ levels within the first postoperative week were recorded (the lowest value was used if multiple measurements were taken on the same day), along with whether the condition improved after corrective interventions, patients were accordingly divided into Low Pa0₂ Group (at least one recorded instance of PaO₂ <80 mmHg) and Normal Pa0₂ Group. Anastomotic leakage was diagnosed based on barium swallow, endoscopy, chest-abdominal CT, or typical clinical signs. By comparing the incidence of anastomotic leakage between the two groups, the relationship between postoperative PaO₂ and anastomotic leakage was analyzed, with further investigation into whether postoperative hypoxemia constitutes an independent and modifiable risk factor.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria required patients diagnosed with esophageal carcinoma or benign esophageal tumors and requiring surgical resection of the lesion with subsequent esophageal reconstruction. Additionally, patients must have had at least one postoperative arterial blood gas analysis and routinely undergone either endoscopy, CT scan, or esophagram for postoperative evaluation of the anastomosis.

Exclusion Criteria:

* We excluded patients who did not require esophageal reconstruction, those undergoing esophageal replacement with colon, and those with incomplete data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective cohort study included patients diagnosed with esophageal carcinoma or benign esophageal tumors who required surgical resection of the lesion followed by esophageal reconstruction. All patients had at least one postoperative arterial blood gas analysis, and anastomotic healing was assessed via esophagram, CT scan, endoscopy, or typical clinical sign.
Sampling Method: Non-Probability Sample
Enrollment: 2083 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Esophageal Anastomotic Leakage Rate | From the date of surgery to 30 days postoperatively
  Anastomotic leak was confirmed by either barium swallow study, CT scan, or endoscopy, or was clinically considered in cases with obvious salivary secretion from the cervical anastomosis.
  The esophageal anastomotic leakage rate was calculated as (the number of patients with a confirmed anastomotic leakage / the total number of patients who underwent esophagectomy) × 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Yang, M.D., Principal Investigator — Department of Thoracic Surgery, Sun Yat-sen University Cancer Center
Locations (1):
- Department of Thoracic Surgery, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided